CLINICAL TRIAL: NCT06469814
Title: Global Registries And Surveys Programme - Heart Failure Snapshot Study (GRASP-HF)
Brief Title: Snapshot Study on Patients With Heart Failure
Acronym: GRASP-HF
Status: Not yet recruiting | Type: Observational
Sponsor: European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: GRASP-HF
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic heart failure
- Patients with acute heart failure

SUMMARY:
The goal of this observational study is to provide a better understanding of medical practice for heart failure management based on real-world data, collected both across Europe and the rest of the world, using robust methodology and representativeness within each country.

Standard management of patients will be the diagnostic and therapeutic interventions routinely performed in each center for patients presenting with signs and symptoms of chronic/acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with chronic or acute Heart Failure (HF), regardless of ejection fraction, either:

• Outpatient with chronic HF (including first-time diagnosis), according to the clinical judgment.

OR

• Patients admitted to hospital or presenting to Emergency Department or Acute out-patient care for acute HF for whom an IV (diuretics, inotropes, vasodilators) or mechanical therapy for HF (mechanical circulatory support) is administered.

Exclusion Criteria:

* Age <18 years
* Patients unwilling to consent (or patient's legally authorized representative unwilling to consent, if the patient is unable to consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all consenting patients seen in the outpatient clinic for chronic HF and all consenting patients admitted for acute HF in the study center as their standard medical care.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to ESC Guidelines in Heart Failure 2021 | 12 months per site
  Full adherence to guidelines for heart failure management

CONTACTS AND LOCATIONS:
Overall Officials: Ovidiu Chioncel, Study Chair — Institute for Cardiovascular Diseases C.C. Iliescu, Bucaresti, Romania

IPD SHARING:
Plan to Share IPD: No